CLINICAL TRIAL: NCT02157636
Title: A Phase 1 Study of CPI-0610, a Small Molecule Inhibitor of BET (Bromodomain and Extra-terminal) Proteins, in Patients With Previously Treated Multiple Myeloma
Brief Title: A Phase 1 Study Evaluating CPI-0610 in Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0610-03
Record Dates: First submitted 2014-05-28; First posted 2014-06-06 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: Phase 1; Oncology; BET Inhibitor
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — CPI-0610

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPI-0610 (Experimental)
  Interventions: Drug: CPI-0610

INTERVENTIONS:
Drug: CPI-0610

SUMMARY:
Open-label, sequential dose escalation and expansion study of CPI-0610 in patients with previously treated multiple myeloma. CPI-0610 is a small molecule inhibitor of bromodomain and extra-terminal (BET) proteins.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥ 18 years)
* Histologically or cytologically confirmed diagnosis of multiple myeloma that has progressed despite at least one line of standard therapy
* Must have measurable disease, defined by one or more of following: (i) a serum M protein > 0.5 g/dl measured by serum protein electrophoresis; (ii) urinary M protein excretion > 200 mg/24 hours; (iii) serum free light chain (FLC) measurement > 10 mg/dl, provided that the serum FLC ratio is abnormal
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate hematological, renal, hepatic, and coagulation laboratory assessments
* Written informed consent to participate in this study before the performance of any study-related procedure

Exclusion Criteria:

* Current infection with HIV, Hepatitis B or Hepatitis C
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of CPI-0610, including any unresolved nausea, vomiting, or diarrhea that is CTCAE grade >1
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * Acute myocardial infarction or angina pectoris ≤ 6 months prior to starting study drug
  * Serum cardiac troponin (cTn) level ≥ 99% percentile of the upper reference limit
  * QTcF > 470 msec on the screening ECG
  * Left ventricular ejection fraction (LVEF) < 50%
* Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded.)
* Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)
* Systemic anti-cancer treatment or radiotherapy less than 2 weeks before the first dose of CPI-0610
* Treatment with an investigational small molecule less than 2 weeks before the first dose of CPI-0610. In addition, the first dose of CPI-0610 should not occur before a period equal to or greater than 5 half-lives of the small molecule investigational agent has elapsed
* Treatment with a therapeutic antibody less than 4 weeks before the first dose of CPI-0610. A minimum 2-week period between the last treatment with a therapeutic antibody and the first dose of CPI-0610 may be permitted in patients with rapidly progressive myeloma, following discussion with the medical monitor
* Treatment with medications that are known to be strong inhibitors or inducers of CYP450 enzymes
* Treatment with medications that are known to carry a risk of Torsades de Pointes
* Immunosuppressive treatment that cannot be discontinued both prior to study entry and for the duration of the study. Oral prednisone at a dose of 10 mg or less per day is allowed, as are other oral corticosteroids given at glucocorticoid-equivalent doses. Topical, nasal and inhaled corticosteroids are also allowed
* Pregnant or lactating women
* Women of child-bearing potential and men with reproductive potential, if they are unwilling to use adequate contraception while on study therapy and for 3 months thereafter
* Patients unwilling or unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLTs) associated with CPI-0610 administration during the first cycle (first 21 days) of treatment | DLTs asessed during Cycle 1 (first 21 days on study)

SECONDARY OUTCOMES:
Safety and tolerability of CPI-0610 as assessed by: frequency of adverse events and serious adverse events; changes in hematology and clinical chemistry values; changes in physical examination, vital signs, electrocardiogram, ECHO and ECOG score | Assessed from Day 1 of Cycle 1 through 30 days after patient's last dose of study drug
Pharmacokinetic parameters of CPI-0610: AUC(0-t), AUC(0-inf), AUCtau,ss, Tmax, Cmax, Ctrough, T1/2, Vd/F, CL/F | Assessed during cycle 1 (first 21 days on study); and on cycle 2, day 1
Pharmacodynamic effects of CPI-0610: Changes in the expression of MYC and other genes in malignant tumor cells; changes in cellular proliferation and in the extent of apoptosis | Assessed during cycle 1 (first 21 days on study); and on cycle 2, day 1
  This outcome measure is a composite measure
Changes in the expression of a set of genes in peripheral blood mononuclear cells (PBMCs) that are sensitive to BET inhibition | Assessed during cycle 1 (first 21 days on study)
Anti-myeloma activity associated with CPI-0610 treatment | Assessed after every cycle of treatment; assessed up to approximately 12 months
  Anti-myeloma activity will be assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma